CLINICAL TRIAL: NCT03621605
Title: A Phase 1 Randomized, Blinded, Placebo-controlled Study to Evaluate the Safety and Tolerability of Single and Multiple Ascending Doses of VIB9600 by Intravenous Infusion or Subcutaneous Injection in Healthy Subjects
Brief Title: A Phase1 Study of VIB9600
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Study terminated due to tolerability issues.
Sponsor: Amgen (Industry)
Collaborators: CTI Clinical Trial and Consulting Services (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Triple | Purpose: Basic Science
Other Study IDs: VIB9600.P1.S1
Record Dates: First submitted 2018-07-18; First posted 2018-08-08 (Actual); Last update posted 2024-12-13 (Actual); Status verified 2024-12

CONDITIONS: Safety Issues

STUDY DESIGN:
Intervention Model Description: A minimum of 56 subjects will be enrolled in 7 planned SAD cohorts (8 subjects per cohort). Subjects enrolled in SAD cohorts will be admitted to a Phase 1 unit and randomized to receive a single dose of VIB9600 or placebo administered by slow IV infusion or SC injection. A minimum of 16 subjects will be enrolled in 2 planned MAD cohorts (8 subjects per cohort). Subjects enrolled in the MAD cohorts will receive VIB9600 or placebo Q2W for 4 weeks (3 doses in total: one each on Days 1, 15 and 29).
Who Masked: Participant, Care Provider, Investigator
Masking Description: Investigator and subject are blinded, sponsor and site pharmacist are unblinded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- VIB9600 (Experimental): Single dose of VIB9600 administered by IV infusion or SC injection.
  Multiple dose VIB9600 administered by IV infusion every 2 weeks for 4 weeks.
  Interventions: Biological: VIB9600
- Placebo (Placebo Comparator): Placebo comparator administered by slow IV infusion or SC injection.
  Interventions: Drug: Placebos

INTERVENTIONS:
Biological: VIB9600 — Part 1 (SAD): IV infusion (30, 100, 200, 300 or 1000 mg) or SC injection (300 mg) on Day 1.
  Part 2 (MAD): IV infusion (100 and 300 mg) every 2 weeks for 4 weeks (3 doses total; Days 1, 15 and 29).
  Arms: VIB9600
Drug: Placebos — Placebo administered by slow IV infusion or SC injection.
  Arms: Placebo

SUMMARY:
Overall design: Single-center, randomized, blinded, placebo-controlled single- and multiple-ascending dose study in healthy adult subjects.

DETAILED DESCRIPTION:
This first-time-in-human (FTIH) SAD and MAD studies in healthy adult subjects will be conducted at one site in the United States of America (USA) on IV and SC VIB9600.

Study acquired from Horizon in 2024. Originally Viela Bio was the sponsor.

ELIGIBILITY:
Key Inclusion Criteria:

1. Healthy male and female subjects aged 18 through 65 years at the time of consent.
2. Body mass index (BMI) of 19.0 through 35.0 kg/m2 at screening and minimum weight of 50 kg.
3. Females must have been surgically sterilized.
4. Nonsterilized male subjects who are sexually active with a female partner of childbearing potential must use a male condom with spermicide from Day 1 through to the final follow-up visit.
5. Able and willing to comply with the requirements of the protocol.

Key Exclusion Criteria:

1. Concurrent enrollment in another clinical study involving an investigational treatment.
2. Received administration of an investigational drug or participated in a device trial within 3 months prior to screening (Visit 1).
3. Subject is a participating investigator, sub-investigator, study coordinator, or employee of the participating site, or is a first-degree relative of the aforementioned.
4. History, or a reason to believe that a subject has a history, of drug or alcohol abuse within the 2 years prior to screening.
5. Positive test for drugs of abuse.
6. Donation of blood or blood products in excess of 500 mL within 3 months prior to screening. Not agreeing to refrain from blood or blood product donations during study participation.
7. Receiving any of the prohibited concomitant medications:

   1. Any immunotherapy or immunosuppressive therapy
   2. Chronic use of steroid medications
   3. Immunoglobulin or blood products
   4. Live vaccines
   5. Anticoagulants
   6. Aspirin

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2018-08-14 (Actual); Primary Completion 2019-04-08 (Actual); Study Completion 2019-04-08 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability of single and multiple doses of VIB9600 | 113 days
  Treatment-emergent adverse events that occur on or after the day of IP administration.

SECONDARY OUTCOMES:
PK of VIB9600 following single- and multiple- dose administration | SAD- Days 1, 2, 3, 5, 8, 16, 29, 43, 57, 85, 113; MAD- Days 1, 3, 8, 15, 22, 29, 32, 36, 43, 57, 86, 113
  Concentration of VIB9600 in serum at different time points after IP administration.
Immunogenicity of VIB9600 following single- and multiple-dose administration. | SAD- Days 1, 15, 29, 57, 85, 113; MAD- Days 1, 15, 29, 57, 85, 113
  Immunogenicity as measured by the presence of anti-drug antibodies (ADA) to VIB9600

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (1):
- CTI Clinical Trial & Consulting Clinical Research Center, Cincinnati, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Jennette JC, Falk RJ, Bacon PA, Basu N, Cid MC, Ferrario F, Flores-Suarez LF, Gross WL, Guillevin L, Hagen EC, Hoffman GS, Jayne DR, Kallenberg CG, Lamprecht P, Langford CA, Luqmani RA, Mahr AD, Matteson EL, Merkel PA, Ozen S, Pusey CD, Rasmussen N, Rees AJ, Scott DG, Specks U, Stone JH, Takahashi K, Watts RA. 2012 revised International Chapel Hill Consensus Conference Nomenclature of Vasculitides. Arthritis Rheum. 2013 Jan;65(1):1-11. doi: 10.1002/art.37715. No abstract available. PMID 23045170
- [Background] Kallenberg CG. Pathogenesis and treatment of ANCA-associated vasculitides. Clin Exp Rheumatol. 2015 Jul-Aug;33(4 Suppl 92):S11-4. Epub 2015 Oct 12. PMID 26457917
- [Background] Kettritz R. How anti-neutrophil cytoplasmic autoantibodies activate neutrophils. Clin Exp Immunol. 2012 Sep;169(3):220-8. doi: 10.1111/j.1365-2249.2012.04615.x. PMID 22861361
- [Background] Ludwig RJ, Vanhoorelbeke K, Leypoldt F, Kaya Z, Bieber K, McLachlan SM, Komorowski L, Luo J, Cabral-Marques O, Hammers CM, Lindstrom JM, Lamprecht P, Fischer A, Riemekasten G, Tersteeg C, Sondermann P, Rapoport B, Wandinger KP, Probst C, El Beidaq A, Schmidt E, Verkman A, Manz RA, Nimmerjahn F. Mechanisms of Autoantibody-Induced Pathology. Front Immunol. 2017 May 31;8:603. doi: 10.3389/fimmu.2017.00603. eCollection 2017. PMID 28620373
- [Background] McKinney EF, Willcocks LC, Broecker V, Smith KG. The immunopathology of ANCA-associated vasculitis. Semin Immunopathol. 2014 Jul;36(4):461-78. doi: 10.1007/s00281-014-0436-6. Epub 2014 Jul 24. PMID 25056155
- [Background] Mulder AH, Heeringa P, Brouwer E, Limburg PC, Kallenberg CG. Activation of granulocytes by anti-neutrophil cytoplasmic antibodies (ANCA): a Fc gamma RII-dependent process. Clin Exp Immunol. 1994 Nov;98(2):270-8. doi: 10.1111/j.1365-2249.1994.tb06137.x. PMID 7955533
- [Background] Nimmerjahn F, Ravetch JV. Anti-inflammatory actions of intravenous immunoglobulin. Annu Rev Immunol. 2008;26:513-33. doi: 10.1146/annurev.immunol.26.021607.090232. PMID 18370923
- [Background] Oganesyan V, Gao C, Shirinian L, Wu H, Dall'Acqua WF. Structural characterization of a human Fc fragment engineered for lack of effector functions. Acta Crystallogr D Biol Crystallogr. 2008 Jun;64(Pt 6):700-4. doi: 10.1107/S0907444908007877. Epub 2008 May 14. PMID 18560159
- [Background] Pagnoux C. Updates in ANCA-associated vasculitis. Eur J Rheumatol. 2016 Sep;3(3):122-133. doi: 10.5152/eurjrheum.2015.0043. Epub 2016 Jan 29. PMID 27733943
- [Background] Porges AJ, Redecha PB, Kimberly WT, Csernok E, Gross WL, Kimberly RP. Anti-neutrophil cytoplasmic antibodies engage and activate human neutrophils via Fc gamma RIIa. J Immunol. 1994 Aug 1;153(3):1271-80. PMID 8027554
- [Background] Sampson HA, Munoz-Furlong A, Campbell RL, Adkinson NF Jr, Bock SA, Branum A, Brown SG, Camargo CA Jr, Cydulka R, Galli SJ, Gidudu J, Gruchalla RS, Harlor AD Jr, Hepner DL, Lewis LM, Lieberman PL, Metcalfe DD, O'Connor R, Muraro A, Rudman A, Schmitt C, Scherrer D, Simons FE, Thomas S, Wood JP, Decker WW. Second symposium on the definition and management of anaphylaxis: summary report--Second National Institute of Allergy and Infectious Disease/Food Allergy and Anaphylaxis Network symposium. J Allergy Clin Immunol. 2006 Feb;117(2):391-7. doi: 10.1016/j.jaci.2005.12.1303. PMID 16461139